CLINICAL TRIAL: NCT06310265
Title: Our Anesthesia Experiment Applied to Child Earthquake Victims in the February 6, 2023 Earthquake
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: TABED 1-24-21
Record Dates: First submitted 2024-02-26; First posted 2024-03-15 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Earthquake; Crush Injury; Anesthesia
Keywords: pediatric; trauma; earthquake; anesthesia
MeSH Terms: conditions — Crush Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective observational study — Our study includes child earthquake victims, regardless of gender, between the ages of 0-18, who applied to our clinic within six months after the February 6, 2023 earthquake and underwent surgery.

SUMMARY:
The study aimed to investigate anesthesia management of pediatric patients in the Ankara Bilkent City Hospital during the earthquake disaster of February 6.

DETAILED DESCRIPTION:
In this study, The investigators planned to retrospectively investigate the anesthesia management of pediatric patients who were transferred to or admitted to the Ankara Bilkent City Hospital in the earthquake disaster of February 6. The anesthesia data on pediatric earthquake victims were insufficient in the literature.The investigators aimed to share our experiences to guide anesthesia management in future possible disasters.

ELIGIBILITY:
Inclusion Criteria:

* Child earthquake victims between the ages of 0-18
* Participants who had surgery and anesthesia between 9 February 2023 and 9 August 2023

Exclusion Criteria:

* The exclusion criterion is child earthquake victims patient who did not undergo anesthesia.

Ages: 30 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: After the earthquake on February 6, pediatric victims were transferred to our hospital and underwent surgery.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-04-05 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
The anesthesia management under pediatric earthquake victims | 6 months (9 February 2023-9 August 2023)
  The effect of general and regional anesthesia practices of Bilkent City Hospital Pediatric Anesthesia practitioners on participant prognosis

CONTACTS AND LOCATIONS:
Overall Officials: Sengul Ozmert, Principal Investigator — Ankara City Hospital Bilkent
Locations (2):
- Turkey (Türkiye) (2):
  - Ankara Bilkent City Hospital, Ankara
  - Ankara Bilkent City Hospital,Department Of Anesthesiology and Reanimation, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozmert S, Isiktekin MD, Taygurt TN, Civelek S, Bayir T, Bayar R, Bostanci SA, Yasar NE. Anesthesia Management of Pediatric Victims After the February 6, 2023, Kahramanmaras Earthquake at a Third-Level Hospital. Paediatr Anaesth. 2025 Nov;35(11):969-976. doi: 10.1111/pan.70039. Epub 2025 Aug 21. PMID 40838437